CLINICAL TRIAL: NCT04259567
Title: Verbesserung Einer gestörten zerebrovaskulären Autoregulation Bei Patienten im Septischen Schock Durch Extrakorporale Reduktion Von Entzündungsmediatoren
Brief Title: Improvement of Cerebrovascular Autoregulation in Patients With Septic Shock Due to Cytokine Elimination
Acronym: SepsAR3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Deputy intensive care unit, Principal investigator, medical doctor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1.0_2019_06_28
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Septic Shock
Keywords: Cerebrovascular Autoregulation; Septic Shock; Cytokine
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filter (Active Comparator): Patients with CytoSorb absorber
  Interventions: Device: Cytokine absorption
- Control (No Intervention): Patients without CytoSorb absorber

INTERVENTIONS:
Device: Cytokine absorption — Use of CytoSorb absorber
  Arms: Filter

SUMMARY:
The trial investigates the effect of cytokine elimination in patients with septic schock and acute renal failure with need for renal replacement therapy on the integrity of cerebrovascular autoregulation. Patients with inclusion criteria were randomly assign in either use of CytoSorb filter integrated in renal replacement therapy versus non additional filter an renal replacement therapy alone. Cerebrovascular autoregulation will be measured with transcranial Doppler ultrasound and correlation with arterial blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* septic shock
* acute renal failure with need for renal replacement therapy

Exclusion Criteria:

* pregnancy
* nursing
* impossibility to do transcranial Doppler ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the index of cerebrovascular autoregulation (Mx) between both groups | days 1 to 4 after diagnosis of septic shock
  Integrity of the cerebrovascular autoregulation will be measured using the index of cerebrovascular autoregulation Mx (moving correlation index). Outcome is the difference of the mean Mx between both groups and, therefore, the difference of integrity of the cerbrovascular autoregulation. A difference of 0.2 in Mx was set as clinically relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of the Johannes Gutenberg-Univerity, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No